CLINICAL TRIAL: NCT01657721
Title: Working Memory Training in Attention-Deficit/Hyperactivity Disorder: Neural Mechanisms of Change
Brief Title: Working Memory Training in ADHD (The Engage Study)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Dr. Rosemary Tannock, Priniciple Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 245899
Record Dates: First submitted 2012-07-27; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Attention-Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wait-list Control (No Intervention): Participants randomized to this group will not undergo The Cogmed Working Memory Training Program during the 5 week period, but will receive weekly phone calls from a member of the research team to review progress and advice on general time management, organization, and mnemonic strategies.
  After a 5-week period, participants in this arm will have access to the working memory training.
- 15 Minute Training (Experimental): Participants will receive a low intensity version of The Cogmed Working Memory Training Program. This involves undergoing 25 training sessions for 15 minutes per day, 5 days a week for 5 weeks. Participants will also receive weekly phone calls from a CogMed Coach to review progress and adjust the training as needed.
  Interventions: Behavioral: Cogmed Working Memory Training Program
- 30 Minute Training (Experimental): Participants will receive the standard-length version of The Cogmed Working Memory Training Program. This involves undergoing 25 training sessions for 30 minutes per day, 5 days a week for 5 weeks. Participants will also receive weekly phone calls from a CogMed Coach to review progress and adjust the training as needed.
  Interventions: Behavioral: Cogmed Working Memory Training Program

INTERVENTIONS:
Behavioral: Cogmed Working Memory Training Program — The Cogmed Working Memory Training Program will be used as the experimental program because of preliminary evidence indicating its effectiveness in enhancing WM and reducing behavioural symptoms of inattention/hyperactivity in children. This software-based training program was designed to improve WM abilities, particularly in children with ADHD or severe attention problems. It includes a set of auditory verbal and visual-spatial WM tasks presented via computer. All tasks involve: maintenance of simultaneous mental representations of multiple stimuli, unique sequencing of stimulus order in each trial and progressive adaptation of difficulty level as a function of individual performance.
  Arms: 15 Minute Training; 30 Minute Training

SUMMARY:
The overall objective of the current study is to determine whether computerized Working Memory (WM) training will enhance WM capacity in college students with Attention Deficit Hyperactivity Disorder (ADHD). There are also four additional objectives. The first is to investigate whether the program's efficacy is impacted by the duration of the daily training sessions. The second is to determine whether improvements in WM will generalize to secondary outcome tasks, such as inhibitory control and planning. The third objective is to examine whether WM training will also ameliorate ADHD symptoms of inattention and hyperactivity. The last objective is to investigate whether improvements will be maintained at a two month follow-up period. The investigators will also be assessing healthy control participants,who will not be receiving treatment, but will be used as a basis of comparison with the ADHD participants,

It is expected that the computerized WM training program will enhance WM capacity in college students with ADHD. In addition, it is believed that these increases in WM capacity will also lead to improvements in other executive functions. It is also hypothesized that WM training will lead to a reduction in ADHD symptomology. Lastly, these improvements should be maintained at three month follow-up.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) and Learning Disability (LD) are among the most common neurobehavioural disorders, with prevalence rates estimated at about 5% to 9% . Approximately 4% of youth in the United States have a comorbid diagnosis of ADHD and a Learning Disability (ADHD/LD). Research has shown ADHD/LD symptoms persist into young adulthood, a time when many are enrolled in post-secondary education. Students with ADHD/LD at the post-secondary education level constitute an emergent subgroup of the ADHD and LD populations that have received far less attention in the literature compared to children, adolescents and employed adults. The actual percentage of college students with ADHD/LD is unknown; however, some estimates suggest that 2-8% of students attending post secondary education have ADHD, LD or both. Youth with the additive problems of both disorders are at high risk for academic failure, and poor psychosocial and occupational outcomes in adulthood. The "multiple deficit model" suggests that there is a common genetic and neuropsychological underpinning to these disorders. For example, ADHD and LD share similar features, such as core deficits in processing speed and working memory. ADHD and LD are each associated with several cognitive difficulties including poor working memory (WM) and processing speed. WM is a "mental workspace" that provides temporary storage and manipulation of information and is closely related to g, a proposed measure of general cognitive ability. In addition, WM has also been found to predict academic achievement. One major problem is that current intervention approaches for ADHD/LD do not target the underlying cognitive deficits fundamental to these diagnoses. Thus, interventions that address underlying cognitive difficulties, such as WM, are a promising avenue of additional treatment for youth with combined ADHD/LD.

WM capacity has generally been thought to be a fixed trait, but recent studies have suggested that it can be improved by intensive and adaptive computerized training. This intervention approach has been evaluated in children and adolescents with ADHD, older adults, and adult stroke patients and shown promising results. Subjects not only improved on the trained WM tasks, but some of the studies suggest that improvements may generalize to non-trained WM activities, complex reasoning tasks, academic functioning, and behavioral symptoms of ADHD or working memory failure. Moreover, brain imaging studies have provided converging evidence of training-related improvements in working memory: specifically increased activation has been found in cortical regions implicated in working memory. However, no studies to date have investigated whether WM capacity can be improved in a population of young adults with ADHD/LD enrolled in post-secondary education programs. Nor have the results been replicated or elaborated upon using different imaging methodologies, like EEG (Electroencephalography), which is able to capture the millisecond time parameters of cognitive processing and so may provide new insights into the neural mechanism of WM and effects of WM training.

The overall objective of the current study is to determine the effectiveness of WM training, as administered by community-based psychologists licensed to provide this training, for college students with ADHD/LD. Specific objectives are to determine whether; i) standard-length computerized WM training enhances WM capacity in college students with ADHD/LD, using behavioral as well as neuro-imaging indices of change; ii) shortened-length WM training would also result in improvements in WM; iii) WM training normalizes WM performance, as compared to typically developing peers (i.e., a healthy comparison group of college students); iv) improvements in WM will generalize to secondary outcome tasks, such as inhibitory control and planning; v) WM training will also ameliorate ADHD symptoms of inattention and hyperactivity; and vi) improvements will be sustained for at least a few months after completing the training.

ELIGIBILITY:
Inclusion Criteria:

* Formal diagnosis of ADHD by a doctor or psychologist
* Registered as a student at a post-secondary institution
* Registered with Student Disability/Accessibility Services at post-secondary institution

Exclusion Criteria:

* Major neurological dysfunction and psychosis
* Current use of sedating or mood altering medication other than stimulants provided for ADHD
* Motor or perceptual handicap that would prevent using the computer program.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Wechsler Adult Intelligence Scale: Digit Span subtest | within 120 days
  This task assesses auditory-verbal working memory. Participants are presented with a series of digits and must immediately repeat them back out loud. If they do this successfully, they are given a longer list.

SECONDARY OUTCOMES:
Adult ADHD Self-Report Scale (ASRS v1.1) | within 120 days
  This instrument consists of eighteen questions based on the criteria used for diagnosing ADHD in adults using DSM-IV-TR criteria.
'Add-3' working memory test | within 120 days
  This task requires participants to add '3' to each digit in a set of 4 digits presented at a constant rate (e.g., the response to the set '3 1 5 4' should be '6 4 8 7')
Cambridge Neuropsychological Testing Automated Battery: Spatial Span Task | within 120 days
  This task presents a set of white squares on a screen, which momentarily change colour in a variable sequence. The participant must then touch the boxes in the same order that they changed colour on the screen. Task demands intensify, as the number of boxes is increased from two to nine. However, if the participant makes an error, the next trial remains at the same difficulty level. Spatial span scores range from 0-9, with the score representing the highest level at which the participant reproduces at least one correct sequence.
Wide Range Assessment of Memory and Learning: Finger-Windows subtest | within 120 days
  This task is a measure of nonverbal, rote sequential recall. The participant is asked to imitate gradually more difficult sequential patterns demonstrated by the examiner.
Barkley Deficits in Executive Functioning Scale (BDEFS) | within 120 days
  This assessment tool evaluates dimensions of adult executive functioning in daily life.
Cognitive Failures Questionnaire | within 120 days
  This self-report questionnaire measures perception, memory, and motor lapses in daily life.
Go-nogo task (N200, P300) | within 120 days
  This task measures response inhibition. The subject is shown sequences of letters and instructed to press a button whenever a letter shows up on the screen, but to withhold a response whenever a letter occurs twice in a row.
Delayed Working Memory Task (P300) | within 120 days
  The participant is shown sequences of either 2 (low load) or 4 (high load) shapes. After a delay period of two seconds, a probe appears and the participant needs to respond by pressing a button whether the probe stimulus was part of the sequence shown before or not.
Selective Working Memory Task (CDA) | within 120 days
  The participant is shown an array of small colored squares to different parts of their visual field. This memory array will consist of either 2 (low load), 4 (high load), or 2 (low load + 2 'distractor' circle) items. After a delay, a test-array is shown and the participant is to respond whether the test-array matched the memory array.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Tannock, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- Ontario Institute of Studies in Education (OISE) at The University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Liu ZX, Glizer D, Tannock R, Woltering S. EEG alpha power during maintenance of information in working memory in adults with ADHD and its plasticity due to working memory training: A randomized controlled trial. Clin Neurophysiol. 2016 Feb;127(2):1307-1320. doi: 10.1016/j.clinph.2015.10.032. Epub 2015 Oct 20. PMID 26541307
- [Derived] Mawjee K, Woltering S, Tannock R. Working Memory Training in Post-Secondary Students with ADHD: A Randomized Controlled Study. PLoS One. 2015 Sep 23;10(9):e0137173. doi: 10.1371/journal.pone.0137173. eCollection 2015. PMID 26397109